CLINICAL TRIAL: NCT03841760
Title: SUV on PSMA PET/CT in Non-Prostate Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollement
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, MD, Chief of Nuclear Medicine, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-1531
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA PET/CT (Experimental): One (1) PSMA PET/CT scan with with either PSMA-11 or DCFPyL
  Interventions: Diagnostic Test: PSMA PET/CT

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT — For 18F-DCFPyL PET/CT: Approximately 9 mCi (333MBq) of 18F-DCFPyL is injected intravenously. Approximately 60-90 minutes following 18F-DCFPyL injection, CT and PET images are consecutively acquired from the base of the skull to the toes.
  For 68Ga-PSMA-11 PET/CT: Approximately 2.5 MBq/kg (0.068 mCi/kg) of 68Ga-PSMA, up to a maximum of 300 MBq (8 mCi), is injected intravenously. Approximately 60 minutes following 68Ga-PSMA injection, CT and PET images are consecutively acquired from the base of the skull to toes.
  Other Names: PSMA PET

SUMMARY:
The objective of this pilot study is to evaluate if 18F-DCFPyL PET/CT or 68Ga-PSMA-11 PET/CT can be used for detection and staging of PSMA-expressing non-prostate tumor.

DETAILED DESCRIPTION:
Prostate specific membrane antigen (PSMA) is a unique membrane bound glycoprotein, which is over-expressed many fold on prostate cancer cells and other types of cancer. Since PSMA is a new target for molecular therapy, PSMA PET/CT allows assessment for therapy in addition to characterization of tumors and staging. Given the success of PSMA PET/CT for prostate cancer and the increasing number of case reports on PSMA uptake in non-prostate cancer, the aim of this project is to fill this literature gap by documenting the avidity of tumors (by means of SUVmax) based on their PSMA immunostaining (by the pathologist) or based on literature report (peer-reviewed article confirming PSMA expression in a tumor type).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older, able to understand and provide written informed consent
* The patient has a tumor known or suspected to have PSMA expression, as reported in the literature or by positive histopathological staining for PSMA.
* The known or suspected tumor must fall into one of the following categories: carcinoma, sarcoma, or hematologic cancer.
* ECOG performance status 0 - 3, inclusive
* Under referring physician's care
* Able to tolerate the physical/logistical requirements of a PET/CT scan including lying supine for up to 40 minutes with the arms above the head and tolerating intravenous cannulation

Exclusion Criteria:

* Patients with neoplasm known in literature to not have PSMA expression, unless patient specific tissue sampling shows PSMA staining on histopathology.
* Medically unstable patients (e.g. acute cardiac or respiratory distress or hypotensive, etc.)
* Patients who exceed the safe weight limit of the PET/CT bed (200 kg) or who cannot fit through the PET/CT bore (70 cm diameter)
* Patients with unmanageable claustrophobia
* Pregnancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Confirm PSMA PET uptake in tumors studied | Immediate
  1. To confirm 18F-DCFPyL PET/CT or 68Ga-PSMA-11 uptake in the known tumor or other lesions found on PSMA PET/CT. The threshold for a positive lesion is a semi-quantitative measurement of activity: SUVmax > 4 in lesions larger than 1.5 cm (so as to offset PET partial volume effect or "camera limitations"). IF SUVmax > 4, the tumor is positive for PSMA PET/CT; If not, the tumor is negative for PSMA PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided